CLINICAL TRIAL: NCT02132065
Title: Unilateral Dual TAP (Transverses Abdominal Plane) Blok i Forbindelse Med Laparoskopisk Nyre Operation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zealand University Hospital (Other)
Responsible Party: Principal Investigator, Nessn Azawi, Consultant, Zealand University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SJ-386
Record Dates: First submitted 2014-05-04; First posted 2014-05-06 (Estimated); Last update posted 2018-01-24 (Actual); Status verified 2018-01

CONDITIONS: Laparoscopic Nephrectomy; TAP Block

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard pain keller (No Intervention)
- TAP block (Experimental): Patients will be scheduled to receive routine analgesic and an unilaterally dual TAP block with 2 points injections of 15 ml of 0,375 % Ropivacain( in total 30 ml 0,375% Ropivacain) in the same side of nephrectomy.
  Interventions: Drug: TAP block

INTERVENTIONS:
Drug: TAP block — Patients will be scheduled to receive routine analgesic and an unilaterally dual TAP block with 2 points injections of 15 ml of 0,375 % Ropivacain( in total 30 ml 0,375% Ropivacain) in the same side of nephrectomy.
  Arms: TAP block

SUMMARY:
Unilaterally Dual TAP (Transversus abdominis plane) block after radical nephrectomy, assessment of benefit and opioid reduction.

Transverses Abdominal Plane (TAP) Block is a relatively new regional technique which infiltrates local anesthetic between the internal oblique and transverse abdominis muscles and provides analgesia to the parietal peritoneum as well as the skin and muscles of the anterior abdominal wall (1). An Ultrasound-guided bilateral dual transversus abdominis plane block (Dual TAP block) had been reported by Boerglum et al (2,3), in which regional anesthesia postoperatively can be provided to the upper (Th6-Th9) and the lower (Th10-Th12) abdominal wall bilaterally using a four-point single-shot technique.

Pain has a wide spectrum of effects on the body. Inadequately controlled postoperative pain may have harmful physiologic, psychological consequences which potentially increase the morbidity and mortality (4,5). It has been recognized that inadequately treated postoperative pain may lead to chronic pain which is often misdiagnosed and neglected (6,7). Chronic postsurgical pain reported in 20% of patients, 6 months after nephrectomy (8).

Hypothesis: The use of unilaterally dual TAP block will reduce the VAS score for pain and the need of morphine postoperatively after radical nephrectomy.

Purpose: To evaluate the analgesic efficacy of unilaterally dual TAP block as an adjuvant to routine analgesic. To assess the difference in morphine usage in the first 48 hours after radical nephrectomy with or without applying of unilaterally dual TAP block.

ELIGIBILITY:
Inclusion Criteria:

-Any patient undergoing laparoscopic nephrectomy- -Age ranges 18-80- -Can read and understand Danish- -Able to give informed consent

Exclusion Criteria:

-History of relevant drug allergy- -Inability to understand written consent forms or give consent- -Age less than 18 or over 80- -Any conversion to open surgery-

-Patients included in ambulant nephrectomy project.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-06; Primary Completion 2017-06 (Actual); Study Completion 2017-06-01 (Actual)

PRIMARY OUTCOMES:
Pain score | 24 hours
  The use of unilaterally dual TAP block will reduce the VAS score for pain and the need of morphine postoperatively after radical nephrectomy

CONTACTS AND LOCATIONS:
Overall Officials: Nessn H. Azawi, MD, Principal Investigator — Roskilde Hospital, Department of Urology
Locations (1):
- Roskilde Hospital, Roskilde, Denmark